CLINICAL TRIAL: NCT05428124
Title: Poor In Vitro Fertilisation Outcomes in Genital Tuberculosis - Case Report
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Kevin Dominique Tjandraprawira, Junior Doctor in Obstetrics and Gynecology, Universitas Padjadjaran
Other Study IDs: OBGY-202206.01
Record Dates: First submitted 2022-06-12; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Tuberculosis, Female Genital; Fertility Disorders
Keywords: In vitro fertilisation; Genital tuberculosis
MeSH Terms: conditions — Tuberculosis, Female Genital | interventions — Fertilization in Vitro; Reproductive Techniques, Assisted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: In vitro fertilisation — In vitro fertilisation
  Other Names: Assisted reproductive technology

SUMMARY:
This is a case series that highlights the challenges in instituting in vitro fertilisation (IVF) treatment amongs genital tuberculosis patients.

DETAILED DESCRIPTION:
In this case series, the investigators recruited patients undergoing IVF treatment previously diagnosed with TB between 01/01/2014 and 30/06/2021. Patients were recruited at the beginning of their IVF treatments. Total sampling was employed for this study.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed genital tuberculosis enrolling in in vitro fertilisation treatment

Exclusion Criteria:

* patients not confirmed to having genital tuberculosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with confirmed genital tuberculosis previously diagnosed during laparoscopy to undergo in vitro fertilisation
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 9 months of gestation
  the number of live births divided by the number of patients recruited

SECONDARY OUTCOMES:
Clinical pregnancy rate | 9 months of gestation
  the number of clinical pregnancies divided by the number of patients recruited

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Tjandraprawirra, M.D., M.Sc., Principal Investigator — Universitas Padjadjaran

IPD SHARING:
Plan to Share IPD: Undecided
anonymised patient data may be shared upon a reasonable written request to the authors team.

REFERENCES:
- [Background] Sharma JB. Current Diagnosis and Management of Female Genital Tuberculosis. J Obstet Gynaecol India. 2015 Dec;65(6):362-71. doi: 10.1007/s13224-015-0780-z. Epub 2015 Oct 7. PMID 26663993
- [Result] Djuwantono T, Permadi W, Septiani L, Faried A, Halim D, Parwati I. Female genital tuberculosis and infertility: serial cases report in Bandung, Indonesia and literature review. BMC Res Notes. 2017 Dec 4;10(1):683. doi: 10.1186/s13104-017-3057-z. PMID 29202851
- [Result] Dai W, Ma L, Cao Y, Wu D, Yu T, Zhai J. In vitro fertilization outcome in women with endometrial tuberculosis and tubal tuberculosis. Gynecol Endocrinol. 2020 Sep;36(9):819-823. doi: 10.1080/09513590.2019.1702639. Epub 2019 Dec 17. PMID 31847626